CLINICAL TRIAL: NCT04661865
Title: Effect of Health Information Package Program (HIP Program) on Knowledge, Compliance , and Hemoglobin Level Among Saudi Pregnant Women With Anemia: A Randomized Controlled Trial
Brief Title: Effect of Health Information Package Program on Knowledge and Compliance Among Pregnant Women With Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Nadia Elsharkawy, Associate Professor - Department of Nursing, College of Applied Medical Sciences, Jouf University, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DSR2020-04-3655
Record Dates: First submitted 2020-11-28; First posted 2020-12-10 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Knowledge; Anemia; Pregnant Women
Keywords: Health Information Package; anemia; pregnant women
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Group A: intervention group who will receive iron supplementation and Heath Information Package Program (HIP program) Group B: Control group: will receive iron supplementation and routine care
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers will interview participants, explain the purpose of the study and they will ask them to sign the consent. All participants will receive iron supplementation and they will learn how to take tablets.
  They will randomly assign in two intervention and control groups (98 each) using a computer-generated table of random numbers and they are unaware of which group they have been assigned to as well as the outcome assessor is unaware
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Routine care only They will receive routine antenatal care that included iron supplementation with follow up of hemoglobin level
  Interventions: Other: Health Information Package Program (HIP program )
- Intervention group (Experimental): They will receive the Heath Information Package Program (HIP program)
  Interventions: Other: Health Information Package Program (HIP program )

INTERVENTIONS:
Other: Health Information Package Program (HIP program ) — Fifteen minutes PowerPoint presentation will be introduced to women to increase women's educational experience and raise their level of engagement and commitment.
  The principal investigator will narrate the video record with PowerPoint slides and it was recorded as a video and will include information regarding the introduction to pregnancy, causes and predisposing factors of iron deficiency anemia during pregnancy, signs and symptoms, prevention, management of iron deficiency anemia during pregnancy that includes iron therapy, iron supplementation, dietary management. Content validity for the information in the video will be done by sending it to three experts in maternity nursing. Iron supplementation will be given to all participants who will start by sixteen weeks of pregnancy and they will receive information regarding the proper usage of iron supplements.

SUMMARY:
Problem description: low compliance with iron supplementation of Saudi pregnant women with anemia is a serious public health concern. The objectives of the study are to determine the effectiveness of the Health Information Package Program (HIP program) in Saudi anemic pregnant women on their compliance with iron supplementation, and level of hemoglobin. Methodology: Randomized Controlled Trial will be conducted on 196 Saudi anemic pregnant women attending the Maternity and Children Hospital in Saudi Arabia their gestational age between 14 and less than 20 weeks. All participants will receive iron supplementation and they will learn how to take tablets. They will randomly assign to two intervention and control groups (98 each) using a computer-generated table of random numbers.

The intervention group will receive a PowerPoint presentation of the Health Information Package Program (HIP program) that will be introduced by the principal investigator, combined with PowerPoint slides to educate women about anemia in pregnancy and send it to them via Whatsapp application while the control group will receive usual care. The participants will be informed about the nature and aim of the study with assuring confidentiality and anonymity. Expected outcome: Health Information Package Program (HIP program) will be effective in terms of increasing women's knowledge regarding anemia during pregnancy, increase compliance with iron supplementation, and hemoglobin level.

DETAILED DESCRIPTION:
The present study aims to assess the efficacy of the Health information package program (HIP program) on compliance with iron supplementation pills, and the level of hemoglobin among Saudi pregnant women with anemia.

The study will be conducted in antenatal outpatient clinics at primary health care centers.

Data Collection tools

I- Demographic and health-related information included data related to women's age, marriage age, level of education, gestational age, parity, body mass index, inter-pregnancy interval, history of excessive or abnormal bleeding during menstruation, and level of hemoglobin.

II- compliance with iron supplementation included questions related to the extent of compliance with iron supplementation among anemic pregnant women and the reason for compliance or non-compliance.

III- The food selection ability checklist contained food items that are rich and poor sources of iron, vitamin C, and protein.

IV- Structured Knowledge Interview Schedule (SKIS): This tool was developed to assess women information before and after the intervention, it contained questions regarding the concept of pregnancy, anemia in pregnancy, causes of iron deficiency anemia, signs and symptoms, the effect of anemia on pregnancy, prevention, and management of iron deficiency anemia. Each correct answer is assigned one point. The maximum number of total possible points was 86.

Random assignment will use to classify the participants equally (98 women each) either in the intervention or control groups using a computer-generated table of random numbers.

ELIGIBILITY:
inclusion criteria

1. Aged between 18-45 years
2. Hemoglobin level less than11 gm/dl and hematocrit less than 30%
3. 14-20 pregnancy weeks
4. Singleton fetus
5. Have a smartphone with internet access (What's App) application
6. Able to read and write
7. Willing to give written informed consent to participate in the study.

Exclusion criteria:

1. Cannot read and write,
2. Have thalassemia or sickle cell anemia.
3. Have a high-risk pregnancy.
4. Had a history of psychiatric illness.
5. Have already started iron supplementation for more than one week.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 1. Aged between 18-45 years
  2. 14-20 pregnancy weeks
  3. pregnant in singleton fetus
Enrollment: 196 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Haemoglobin | after three months ( 90 days ± 7 days)
  > 11 gm/ dl

SECONDARY OUTCOMES:
knowledge | after three months ( 90 days ± 7 days) - study period
  The overall number of knowledge related questions is 86 High knowledge: 57-71 Moderate knowledge: 36- 56 tablets Low knowledge: <36 tablets
compliance with iron supplementation | after three months ( 90 days ± 7 days)
  The overall number of iron tablets that should have been taken during the three month study period will be 90
  High compliance: 68-90 tablets Moderate compliance: 45- 67 tablets Low compliance: <45 tablets

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Health Care centers, Jouf- Saudi Arabia, Jouf, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
1. No personal identification data will be collected, so the researchers assure participants' anonymity.
  2. The researchers will collect only the data required to this study.
  3. Demographic data of participants will be coded to maintain confidentiality.
  4. All submitted data are saved and handled electronically by the researchers only through password-protected files.